CLINICAL TRIAL: NCT01243346
Title: Phase II Study of Crenolanib (CP-868,596), a Selective and Potent Inhibitor of PDGFR, for the Treatment of Patients With Advanced Gastrointestinal Stromal Tumors With the D842-related Mutations and Deletions, Including the D842V Mutation, in the PDGFRA Gene
Brief Title: Study of Crenolanib for the Treatment of Patients With Advanced GIST With the D842-related Mutations and Deletions in the PDGFRA Gene
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARO-BRE-002
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: D842-related Mutant GIST
Keywords: Gastrointestinal Stromal Tumor; PDGFR Inhibitor; Crenolanib (CP-868,596)
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Crenolanib (CP-868,596) (Experimental)
  Interventions: Drug: Crenolanib besylate (CP-868,596-26), Dose: 140mg BID

INTERVENTIONS:
Drug: Crenolanib besylate (CP-868,596-26), Dose: 140mg BID — Highly potent inhibitor of both PDGFR receptors alpha and beta

SUMMARY:
This Phase II study is designed to evaluate the antitumor efficacy and pharmacokinetics of crenolanib (CP-868,596) in patients with D842-related mutant metastatic GIST.

DETAILED DESCRIPTION:
Crenolanib (CP-868,596) is an orally bioavailable, selective inhibitor of PDGFR receptor tyrosine kinase with IC50s of 0.4 ng/mL and 0.8 ng/mL for PDGFRα and PDGFRβ, respectively.

In preclinical models of cell lines with the D842V mutation in the PDGFRA gene, crenolanib (CP-868,596) blocked phosphorylation of PDGFRα at nanomolar concentrations, suggesting that it may provide a clinical benefit to patients with D842V mutant GIST.

In addition, crenolanib was also active in inhibiting phosphorylation of cell lines with two point mutations (double mutants) PDGFRA V561D + D842V and PDGFRA T674I + D842V.

ELIGIBILITY:
Inclusion Criteria

* Male or female, of any racial or ethnic group
* Age 18 years or older
* Life expectancy of greater than 12 weeks
* Patient able and willing to provide informed consent
* Normal liver function, defined as AST and ALT ≤2.5x ULN, and Total Bilirubin ≤ 2x ULN.
* Total creatinine ≤ 1.5x ULN
* ECOG Performance Status 0 - 2 (Appendix II)
* Patients must have histologically or cytologically confirmed GIST with a D842-related mutation or deletion on the PDGFRA gene
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See Section 10.1.2 for the evaluation of measurable disease.
* Patients must have recovered from any prior therapy and completed the minimum of, either 5 half-lives of prior therapy or 2 weeks must have elapsed since prior treatment

Exclusion Criteria

* Patient unable to provide informed consent
* ECOG Performance status > 2
* Any concurrent anticancer therapy, immunotherapy, or hormonal therapy.
* Any other investigational agents taken within 2 weeks of start of study drug or if study drug will commence within 5 half-lives of prior therapy
* Patients with known or active Hepatitis B or C; liver cirrhosis.
* Patients with active fungal, viral, and bacterial infections
* Positive serum pregnancy test
* Pregnant or lactating women
* Patients on concomitant medications that induce or inhibit CYP3A4 (Appendix III)
* Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol e.g. impairment of gastrointestinal (GI) function, or GI disease that may significantly alter the absorption of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The primary end-point is overall response rate | 1.5 years
  To determine the response rate of patients with advanced D842V mutant GIST, when treated with Crenolanib (CP-868,596). Response will primarily be determined by RECIST criteria

SECONDARY OUTCOMES:
Progression free survival rate | 6 months
  To determine the progression free survival rate at 6 months in patients with advanced GIST with the D842V mutation in the PDGFRA gene, when treated with CP-868,596 (crenolanib).
Obtain toxicity information | 1 year
  To obtain additional toxicity information in patients with advanced GIST with the D842V mutation in the PDGFRA gene.
PKPD analysis | 1 year
  To obtain additional PK, pharmacodynamic and plasma inhibitory assay information in patients with advanced GIST with the D842V mutation in the PDGFRA gene.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret von Mehren, MD, Principal Investigator — Fox Chase Cancer Center; Michael C Heinrich, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Knight Cancer Institute, Oregon Health and Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Heinrich MC, Griffith D, McKinley A, Patterson J, Presnell A, Ramachandran A, Debiec-Rychter M. Crenolanib inhibits the drug-resistant PDGFRA D842V mutation associated with imatinib-resistant gastrointestinal stromal tumors. Clin Cancer Res. 2012 Aug 15;18(16):4375-84. doi: 10.1158/1078-0432.CCR-12-0625. Epub 2012 Jun 27. PMID 22745105
- See also: Fox Chase Cancer Center — http://www.fccc.edu
- See also: OHSU Knight Cancer Institute — http://www.ohsu.edu/xd/health/services/cancer/